CLINICAL TRIAL: NCT00588510
Title: Detection of Circulating Osteosarcoma Tumor Cells in the Blood of Patients Using the Polymerase Chain Reaction
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 99-120
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Osteosarcoma
Keywords: Sarcoma; Bone
MeSH Terms: conditions — Osteosarcoma; Sarcoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood draw: Peripheral blood samples (6-9 ml) will be collected in purple top tubes, when routine laboratory tests are being drawn. The blood will be drawn through central venous catheters, whenever possible.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Peripheral blood samples (6-9 ml) will be collected in purple top tubes, when routine laboratory tests are being drawn. The blood will be drawn through central venous catheters, whenever possible. Blood will be drawn once from patients with malignant diagnoses other than osteosarcoma, neuroblastoma, Ewing's sarcoma or synovial sarcoma. In patients with osteosarcoma we will obtain blood when baseline laboratory tests are obtained, after every two cycles of treatment (approximately every six weeks), at the end of planned surgery and chemotherapy, every three months for the first year off therapy and yearly thereafter. We will also obtain blood if the patient relapses.

SUMMARY:
This study focusses on finding out if osteosarcoma can be detected in blood. The cells will be measured by a new laboratory technique called the polymerase chain reaction. This new technique can identify one tumor cell among one million normal cells. Using this technique Memorial Sloan-Kettering Cancer Center research doctors may be able to detect tumor cells that could not be identified any other way. This test will be in addition to cancer treatment and will not replace any other test used normally. As this technique is still unproved the results will not be given to patients or patient's doctors and will not be used to change cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteosarcoma are the study group
* Patients with malignant diagnoses other than osteosarcoma, neuroblastoma, Ewing's sarcoma or synovial sarcoma may participate as controls
* Histologically proven osteosarcoma or a history of histologically proven osteosarcoma are eligible for participation. The patient does not need to be newly diagnosed for enrollment on this protocol
* Patients with malignant diagnosis other than osteosarcoma, neuroblastoma, Ewing's sarcoma or synovial sarcoma are eligible to participate if they have a central venous catheter and routine blood work is being drawn

Exclusion Criteria:

* Patients less then three years of age
* Patients with Ewing's sarcoma, neuroblastoma and synovial sarcoma will be excluded from this protocol

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Osteosarcoma patients seen in the Pediatrics Department or the Orthopedic Division of the Surgery Department at Memorial Sloan-Kettering Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2000-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine if circulating osteosarcoma cells can be reliably detected and quantitated in the blood of patients with localized and advanced osteosarcoma. | conclusion of the study

SECONDARY OUTCOMES:
To determine the frequency circulating osteosarcoma cells can be detected in the blood of patients at diagnosis, during therapy, at the completion of all planned therapy and at relapse. | conclusion of the study
To determine if the presence of circulating osteosarcoma tumor cells is associated with patient outcome. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Paul Meyers, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm